CLINICAL TRIAL: NCT06121765
Title: Metabolic Alternation and Clinicohematological Characteristic in Chronic Phase CML in Patient Treated With TKI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Rabea Abdelrahman Soltan, Principal investigator, Assiut University
Other Study IDs: Metabolic alteration in CML
Record Dates: First submitted 2023-10-29; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: CML, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Tyrosine Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tyrosine kinase inhibitor — Follow up base metabolic index,lipid profile, HbA1c, thyroid function in CML patients treated with TKI

SUMMARY:
Metabolic alternation and clinicohematological characteristic in chronic phase CML in patient treated with TKI

DETAILED DESCRIPTION:
Chronic myeloid leukemia (CML), a clonal hematopoietic stem cell malignancy, is characterized by unique translocation leading to the formation of the Philadelphia chromo- some.Because of the specific genotype knowledge, tyrosine kinase inhibitors have been used in CML and have significantly improved the prognosis of patients with CML, especially n high-income countries like the United States.Notably, the 5-year survival rates increased from 40% to 90%. So, CML is increasingly seen as a chronic instead of a potentially fatal disease.

Obesity is increasingly prevalent worldwide and is considered o be an important risk factor for adverse outcomes in many cancers.

Obesity is well-known for being associated with metabolic abnormalities like hyperglycemia, hypertension, or dyslipidemia.The metabolic abnormalities and obesity- induced systemic chronic inflammation contribute to tumorigenesis and progression.

Obesity alone may not reflect the actual metabolic health state, and it appears to be more accurate to reclassify patients based on the combination of body mass index (BMI) and metabolic status to further determine the relationship between obesity itself or the combination of metabolic status and prognosis of patients with CML.

Triglyceride-to-high-density lipoprotein cholesterol ratio (TG/HDL-C) has been proposed as a reliable and simple alternative to assess atherogenic index, insulin resistance, and dyslipidemia.[8] Furthermore, positive relationships between the TG/HDL-C ratio and various clinical features of many cancers, such as tumor stage and tumor type, have been reported in previous studies.[9] These findings warrant further studies to explore TG/ HDL-C ratio with respect to TKI administration in CML and as a factor associated with side effects, and potentially, to assess its role in prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient newly diagnosed with CML and received TKI

Exclusion Criteria:

* patient previously diagnosed CML and started treatment or in post treatment follow up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic myeloid leukemia (CML), a clonal hematopoietic stem cell malignancy, is characterized by unique translocation leading to the formation of the Philadelphia chromo- some.1 Because of the specific genotype knowledge, tyrosine kinase inhibitors have been used in CML and have significantly improved the prognosis of patients with CML, especially n high-income countries like the United States.2,3 Notably, the 5-year survival rates increased from 40% to 90%. So, CML is increasingly seen as a chronic instead of a potentially fatal disease.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of BMI in patient diagnosed CMLm b. S Evaluat BMI in patient newly diagnosed CMLm , Triglyceride-to-High Density Lipoprotein Cholesterol Ratio b. S | Base line
  Evaluation of weight in kg and height in meter will be combined to measure BMI in (kg/m2)